CLINICAL TRIAL: NCT07118384
Title: Comparison of the Clinical Efficacy of Ampicillin/Sulbactam and Cefoperazone/Sulbactam Against Multidrug Resistant Acinetobacter Baumannii Infections in Critically Ill Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayah Mohammed Khalil Ibrahem, Senior Clinical pharmacist -Trauma and surgical ICU ER185 at Kasr alainy hospital, MSc , BCPS, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-138-2025
Record Dates: First submitted 2025-06-20; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Acinetobacter Baumannii Infection
Keywords: Acinetobacter baumannii; cefoperazone- sulbactam; ampicillin-sulbactam
MeSH Terms: interventions — sultamicillin

STUDY DESIGN:
Intervention Model Description: Open-labeled, Parallel, Randomized, Controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ampicillin- sulbactam (Active Comparator): Intravenous ampicillin-sulbactam (2:1)
  Interventions: Drug: Ampicillin - Sulbactam Injection
- Cefoperazone-sulbactam (Experimental): intravenous cefoperazone-sulbactam (1:1)
  Interventions: Drug: Cefoperazone-sulbactam injection

INTERVENTIONS:
Drug: Cefoperazone-sulbactam injection — Two grams of Cefoperazone/sulbactam IV are administered every 8 hours, and each dose is administered as an extended infusion over 4 hours. The solution is diluted with a compatible solution (normal saline 0.9%) with a maximum final concentration of 250 mg/ml
  Arms: Cefoperazone-sulbactam
Drug: Ampicillin - Sulbactam Injection — Two grams of Ampicillin/sulbactam IV are administered every 8 hours, and each dose is administered as an extended infusion over 4 hours. The solution is diluted with a compatible solution (normal saline 0.9%) with a final concentration not exceeding 45mg/ml.
  Arms: Ampicillin- sulbactam

SUMMARY:
To compare the clinical effectiveness of two different sulbactam-based regimens (ampicillin-sulbactam versus cefoperazone-sulbactam) in the treatment of Acinetobacter baumannii infections in critically ill patients.

DETAILED DESCRIPTION:
Among Acinetobacter species, Acinetobacter baumannii is the most important member and is commonly implicated in nosocomial infections. Acinetobacter baumannii is a gram-negative coccobacillus that has emerged from an organism of questionable pathogenicity to an infectious agent of importance to hospitals worldwide. In the intensive care unit ICU setting, Acinetobacter baumannii has been implicated in severe and occasionally life-threatening infections such as ventilator-associated pneumonia and bloodstream infections. Acinetobacter baumannii can produce biofilms in environments exposed to antibiotics; thus, it can survive for long periods and easily develop multidrug (MD), extremely or extensively drug (XD), and even pan-drug resistances (R) to various types of antibiotics, resulting in high patient mortality.

The underlying mechanisms can be divided into three categories. First, A. baumannii produces decomposition enzymes that deactivate antibiotics. Second, it can reduce or hinder the entry of antibiotics. For example, A. baumannii prevents the entry of antibiotics by controlling efflux pumps, or it can remove the antibiotics that have entered the cells. Third, point mutations alter the targets or functions of bacteria and reduce their affinity for antibiotics. Owing to its strong infectivity and drug resistance, A. baumannii has been added to the list of the World Health Organization's antibiotic-resistance priority pathogens.

Sulbactam, a beta-lactamase inhibitor, is commercially available mainly in combination with β-lactam antibiotics (as in ampicillin-sulbactam or cefoperazone-sulbactam), is a drug containing a beta-lactam ring derived from 6-aminopenicllanic acid. It can bind to the active sites of b-lactamase antibiotics to protect against antibiotic hydrolysis and restore antibiotic activity.

The antimicrobial property distinguishing sulbactam from other beta-lactamase inhibitors is its activity against Acinetobacter spp. Therefore, sulbactam is an alternative treatment option due to the worldwide spread of multidrug resistance Acinetobacter baumannii, for which only a few effective antimicrobial agents are currently available. The Infectious Diseases Society of America Antimicrobial-Resistant Treatment Guidance suggests that high-dose ampicillin-sulbactam (total daily dose of 6-9 grams of the sulbactam component) be included in the combination therapy regimen. If ampicillin-sulbactam non-susceptibility is shown, high-dose ampicillin-sulbactam can still be a helpful therapy choice. Acinetobacter baumannii isolates in China were more susceptible to cefoperazone-sulbactam than to ampicillin-sulbactam (resistance rates 48.8% vs 59.1%). The literature's limited data indicated that patients with Acinetobacter baumannii may expect moderate clinical benefits with Cefoperazone -Sulbactam. Salvation therapy may be attempted with combination treatment, particularly with polymyxins. There are no randomized controlled studies investigating the effectiveness of cefoperazone-sulbactam in the presence or absence of polymyxins for Acinetobacter baumannii infections.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. Age ≥21 years old.
  2. Patient with signs and symptoms of sepsis.
  3. positive culture Carbapenem-resistant Acinetobacter baumannii (CRAB).

Exclusion Criteria:

* Exclusion criteria:

  1. Empirical sulbactam-based therapy against Gram-negative bacteria
  2. History of hypersensitivity reactions to ampicillin-sulbactam/cefoperazone-sulbactam

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Treatment effectiveness Based on Clinical improvement | 5 days
  Clinical response will be assessed by ICU physicians based on physical examination findings and daily clinical records on Day 5 of treatment.
  Patients will be classified into one of the following categories:
  * Cure: Complete resolution of signs and symptoms related to the infection
  * Failure: No improvement, persistence of symptoms beyond 72 hours, or deterioration requiring antibiotic escalation Unit of Measure: % of patients with clinical cure or failure Clinical evaluation performed daily by ICU physicians using physical examination and patient records, in accordance with standardized definitions of clinical response outlined by the CDC (Centers for Disease Control and Prevention) and IDSA (Infectious Diseases Society of America) 2024-2025 guidelines including primary blood stream infection-skin and soft tissue and surgical site infection-intra abdominal infection- lower respiratory infection- urinary tract infection- catheter related infection and bone and joint infection.

SECONDARY OUTCOMES:
Bacteriological Response Assessed by Culture and Sensitivity Testing | 5 days
  Microbiological eradication will be assessed using microbiological cultures collected on Day 5 from appropriate clinical specimens (e.g., sputum, blood, wound, urine, central line ).
  Categories of response include:
  * Eradication: No growth of Acinetobacter baumannii
  * Persistence: Continued growth of A. baumannii
  * Superinfection: Growth of a new microorganism Unit of Measure: % of patients with eradication, persistence, or superinfection Antimicrobial susceptibility of the isolated bacteria was determined by the Kirby-Bauer disc diffusion method based on the Clinical and Laboratory Standard Institute (CLSI) guideline. The isolates resistant to 2 or more drug classes simultaneously were considered to be multidrug resistant (MDR) (hospital microbiology laboratory).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Mukhtar, Professor Anesthesia and ICU, Study Director — Cairo Univesrsity hospitals Kasr Alainy
Locations (1):
- Cairo university hospitals kasr alainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided